CLINICAL TRIAL: NCT03176485
Title: Pilot Study to Evaluate the Signaling Pathway Modulation Demonstrated by Raf, MEK, and Kinase Inhibitors In Human Skin With or Without Solar Simulated Light
Brief Title: Evaluation of Pathway Modulation by Raf, MEK, & Kinase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1409505107
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Cancer; Melanoma; Colon Cancer; Differentiated Thyroid Cancer; Hepatocellular Carcinoma; Renal Cell Carcinoma; Metastatic Melanoma; HCC; Metastatic Colon Cancer
Keywords: metastatic; melanoma; cancer; colon; thyroid; Differentiated; Hepatocellular Carcinoma; HCC; RCC; Renal Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Colonic Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Neoplasms; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ArmA: With Solar Simulated Light Exposure (Experimental)
  Interventions: Other: Solar Simulator
- ArmB: With Solar Simulated Light Exposure (Vemurafenib/Dabraf) (Experimental): Subjects in this study arm undergo the same procedures as Arm A, with the addition of a blood test for the presence of porphyrins
  Interventions: Other: Solar Simulator
- ArmC: Without Solar Simulated Light Exposure (No Intervention)

INTERVENTIONS:
Other: Solar Simulator — A Multiport UV Solar Simulator Model 600 (Solar Light Co., Inc., Philadelphia, PA) will be used to administer Solar Simulated Light (SSL) exposures to formerly unexposed buttock skin.The device is equipped with six 8mm liquid light guides (LLG), allowing for 6 simultaneously conducted exposures.A large 3x2 endplate places the LLGs several centimeters apart and is specifically designed for Sun Protection Factor (SPF) and photo patch testing. The dose of emission from each LLG can be precisely regulated and the spectrum of emission can be limited to UVA (320-390 nm) or UVB+UVA (290-390 nm). The operator can select between UVA only and a combined Ultraviolet-A (UVA)/ Ultraviolet-B (UVB) spectrum by placement of an optical filter. The spectral output (indicated below) follows the distribution of sunlight from 290 to 390 nm.
  Other Names: Multiport UV Solar Simulator Model 60
  Arms: ArmA: With Solar Simulated Light Exposure; ArmB: With Solar Simulated Light Exposure (Vemurafenib/Dabraf)

SUMMARY:
This is a pilot study designed to evaluate the cutaneous effect of systemic inhibition of the tyrosine kinase pathway in the presence or absence of solar simulated light exposure.

A maximum of 45 subjects will be accrued into the overall study we anticipate approximately 25 patients in the Raf inhibitor group and 10 patients each into the Tyrosine Kinase and MEK inhibitor arms of the study.

DETAILED DESCRIPTION:
The study will evaluate the modulatory effect of systemic Raf inhibition in the MEK/ERK and PI3 /Akt/mTOR pathways in patients undergoing targeted therapy for metastatic disease.

Changes in relevant proteins will be evaluated using a combined protein expression methodology that in includes immunohistochemistry (IHC) and reverse phase protein microarray (RPPA) technology.

The primary endpoint of this study will be assessed in normal skin and skin acutely exposed to solar simulated light

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have not yet initiated but plan to undergo dosing with a Tyrosine Kinase inhibitor (TKI) or Raf inhibitor, either alone or with a MEK inhibitor, for treatment of metastatic melanoma, colon cancer, hepatic cell carcinoma, or thyroid cancer.
* Individuals with normal skin and Fitzpatrick skin type II, III or IV.
* Individuals who are willing to limit sun exposure to the body during the study period, and who agree to wear protective clothing and SPF 50 broad spectrum sunscreen or sunblock on exposed skin when they are outdoors.
* Individuals who have the ability to understand and willingness to sign an informed consent before initiation of study procedures, after the nature of the study is explained to them and they have asked any questions.
* Individuals with a Karnofsky Performance Status of at least 80%.

Exclusion Criteria:

* Individuals with any inflammation or irritation of the skin at the test area (buttocks), or any skin conditions felt by the study physician to contraindicate enrollment.
* Individuals with a history of any skin cancer, melanocytic lesions, actinic keratoses or actinic damage in the test area are ineligible. History of such conditions at a body site other than the test area is not exclusionary if in the opinion of the study physician it will not pose a risk to the subject.
* Individuals who are immunosuppressed by virtue of medication or disease, as determined by the examining study physician. This includes AIDS patients and subjects taking oral steroids.
* Individuals with active infection, psychiatric illness, or other situations that in the opinion of the study physician limit compliance or interfere with the study regimen.
* Individuals with a history of photosensitive diseases including, but not limited to, Lupus Erythematosus, pseudoporphyria, or other diseases that in the opinion of the study physician would pose a risk to the subject or interfere with the study.
* Individuals who have used photosensitizing drugs within the last 30 days prior to study enrollment, or who will be using a photosensitizing drug during the time of the study.
* Individuals who have used any topical medication other than emollients on the test area within 30 days prior to study enrollment.
* Individuals who have used retinoids, steroids, 5-fluorouracil, Levulan, Vaniqua (eflornithine), Solaraze, or Imiquimod (Aldara®) anywhere on the body within 30 days prior to enrollment.
* Individuals must not take mega-doses of vitamins. Mega-doses are defined as more than 5 capsules of standard multivitamins daily or more than the Tolerable Upper Intake Levels of Vitamins, as defined by the Institute of Medicine, National Academy of Sciences. Such vitamin therapy must be discontinued at least 30 days prior to study entry.
* Individuals with a history of natural or artificial sun exposure to the buttocks within 30 days of study participation.
* Individuals with Fitzpatrick skin type I
* Individuals with Fitzpatrick skin type V or VI
* Individuals enrolled in or who plan to enroll in a clinical intervention trial. There must be a 30-day period between completing a previous study and enrolling in this study. The Principal Investigator will have the option to consider an exception for patients on drugs of interest for the purpose of this study.
* Individuals with a known allergy to lidocaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-10-17 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Modulatory effect of systemic Raf inhibition in the MEK/Erk and PI3 /AKT/mTOR pathways in patients undergoing targeted therapy for metastatic disease | 2 months
  The primary endpoint of the study is to evaluate the modulatory effect of systemic Raf inhibition in the MEK/Erk and PI3 /AKT/mTOR pathways in patients undergoing targeted therapy for metastatic disease. Changes in relevant proteins will be evaluated using a combined protein expression methodology that in includes immunohistochemistry (IHC) and reverse phase protein microarray (RPPA) technology. The primary endpoint of this study will be assessed in normal skin and skin acutely exposed to solar simulated light.

SECONDARY OUTCOMES:
Downstream modulation of direct Ras and MEK inhibition in human keratinocytes and melanocytes following acute solar simulated light exposure in the presence of metastatic disease treatment with Tyrosine kinase and MEK inhibitors. | 2 months
  The modulatory effect will be evaluated using IHC and RPPA technology.
Modulatory effect of systemic Raf inhibition in the MEK/Erk and PI3 /AKT/mTOR pathways in eligible melanocytic nevi. | 2 months
Correlate the type and severity of cutaneous squamous cell carcinoma development in patients treated with BRaf inhibitors and the modulatory profile identified in the proposed primary endpoint. | 2 months
Safety of performing solar simulated light studies in patients undergoing Ras inhibition for metastatic disease. | 2 months
Modulatory effect of Ras inhibition in Epidermal Growth Factor Receptor (EGFR) and Activating Protein-1 (AP1) signaling pathways (IHC and RPPA). | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel-Lewandroski, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided